CLINICAL TRIAL: NCT00796263
Title: Antiretroviral Therapy for Acute and Chronic HIV Infection
Acronym: AAHIV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Somchai Sriplienchan, MD, Executive Director of SEARCH Research Foundation, SEARCH Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAART for Acute HIV infection
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Acute HIV Infection; Chronic HIV Infection
Keywords: Acute HIV infection; Chronic HIV infection
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAART (Other): The proposed HAART regimen consists of:
  * 1 or 2 nucleoside/nucleotide analog reverse-transcriptase inhibitor (NRTI) class medications plus
  * Dolutegravir(DTG) 50 mg orally once daily
  Interventions: Drug: HAART

INTERVENTIONS:
Drug: HAART — 1 (lamivudine) or 2 (lamivudine + abacavir) nuceloside/nucleotide analog reverse-transcriptase inhibitor (NRTI) class medications once daily
  plus
  dolutegravir(DTG) 50 mg orally once daily
  Other Names: Triumeq; Dovato

SUMMARY:
The purpose for this protocol is to provide safe and effective standard ART to SEARCH 010 and SEARCH 013 participants. Participants are enrolled in an acute HIV infection study (SEARCH 010 protocol: 'Establish and characterize an acute HIV infection cohort in a Thai high-risk population') or in a study of chronic HIV infection (SEARCH 013 protocol 'Characteristics of immunity in gut mucosa, spinal fluid, lymph node and blood of HIV negative and HIV positive Thais').

DETAILED DESCRIPTION:
To compare systemic and tissue compartments (genital secretion, CNS, gut and lymph node) outcomes among individuals who initiate HIV treatment during acute vs. chronic HIV infection. The outcomes will be compared by stages of infection and antiretroviral regimens. Participants are enrolled in an acute HIV infection study (SEARCH 010 protocol: 'Establish and characterize an acute HIV infection cohort in a Thai high-risk population') or in a study of chronic HIV infection (SEARCH 013 protocol 'Characteristics of immunity in gut mucosa, spinal fluid, lymph node and blood of HIV negative and HIV positive Thais') with the latter serving as controls for the acutely infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Enrolled in the SEARCH 010 or 013 protocols with documentation of acute or chronic protocol defined HIV-1 infection and chooses to initiate or continue ART
3. Understand the study and sign informed consent form. Persons who cannot read will have the consent form read and explained to them by a member of the study staff and they can give informed consent by using their thumb print
4. Availability for follow-up for the planned study duration

Exclusion Criteria:

1. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2009-05-13 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
HIV-related clinical events | 10 years
Immunologic parameters including CD4 count and CD4/CD8 ratio | 10 years
Virologic parameters including HIV RNA and HIV reservoir markers | 10 years

SECONDARY OUTCOMES:
Adverse events related to HAART initiated during acute HIV infection as assessed by DAIDS grading table version 2.1 | 10 years
Adherence to ART | 10 years
Frequency and functional status of HIV-specific CD8+ T cells in blood and tissue compartments (genital secretion, CSF, gut and lymph node) | 10 years
Expression of non-specific activation markers on CD8+ T cells in blood and tissue compartments (genital secretion, CSF, gut and lymph node) | 10 years
HIV drug resistance by genotyping at study baseline and in case of virological failure after viral suppression. | 10 years
Assessment of immune activation markers by multiplex technology in blood plasma, CSF and colon and lymph node cell suspension | 10 years
Determination of Z-score of 4 neuropsychological tests of motor and processing speed, the so-called NPZ4 score. | 10 years
  The NPZ-4 score, a composite score of neuropsychological testing ranges from -2.2 to 2.1, with a mean of 0. The score is used to assess cognitive function in studies involving HIV and antiretroviral therapy. A higher score indicates better cognitive performance.
Assessment of functional brain magnetic resonance imaging and magnetic resonance spectroscopy | 10 years
Assessment of impact of co-morbid infections on CD4 count, CD4/CD8 ratio and HIV VL | 10 years
  The impact of syphilis and COVID-19 on CD4 count, CD4/CD8 ratio and HIV VL will be assessed during co-infection and after resolution. Given the duration of cohort follow-up, additional or new infections may be assessed for impact as incidence in the cohort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Somchai Sriplienchan, MD, MPH, Principal Investigator — SEARCH Research Foundation
Locations (1):
- Institute of HIV Research and Innovation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ananworanich J, Eller LA, Pinyakorn S, Kroon E, Sriplenchan S, Fletcher JL, Suttichom D, Bryant C, Trichavaroj R, Dawson P, Michael N, Phanuphak N, Robb ML. Viral kinetics in untreated versus treated acute HIV infection in prospective cohort studies in Thailand. J Int AIDS Soc. 2017 Jun 26;20(1):21652. doi: 10.7448/IAS.20.1.21652. PMID 28691436
- [Derived] de Souza MS, Pinyakorn S, Akapirat S, Pattanachaiwit S, Fletcher JL, Chomchey N, Kroon ED, Ubolyam S, Michael NL, Robb ML, Phanuphak P, Kim JH, Phanuphak N, Ananworanich J; RV254/SEARCH010 Study Group. Initiation of Antiretroviral Therapy During Acute HIV-1 Infection Leads to a High Rate of Nonreactive HIV Serology. Clin Infect Dis. 2016 Aug 15;63(4):555-61. doi: 10.1093/cid/ciw365. Epub 2016 Jun 17. PMID 27317797